CLINICAL TRIAL: NCT02173132
Title: Acetyl-L-Carnitine Reduces Perceived Work Stress and Improves Work Ability and Work Performance in Hepatic Encephalopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/2010
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Work Stress; Work Ability; Work Performance
MeSH Terms: conditions — Occupational Stress | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- acetyl-L-carnitine (Active Comparator): 2 g acetyl-L carnitine twice a day for 90 days
  Interventions: Drug: Acetyl-L-carnitine
- sugar pill (Placebo Comparator): Placebo twice a day for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetyl-L-carnitine
  Arms: acetyl-L-carnitine
Other: Placebo
  Arms: sugar pill

SUMMARY:
This study evaluated the effects of acetyl-L-carnitine treatment on Perceived Work Stress, Work Ability and Work Performance in subjects with Hepatic Encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* overt hepatic encephalopathy (HE) or a history of overt HE

Exclusion Criteria:

* history of recent alcohol intake; infection; recent antibiotic use or gastrointestinal bleeding; history of recent use of drugs affecting psychometric performances like benzodiazepines, antiepileptics or psychotropic drugs; a history of shunt surgery or transjugular intrahepatic portosystemic shunt for portal hypertension; electrolyte imbalance; renal impairment; hepatocellular carcinoma; severe medical problems such as congestive heart failure, pulmonary disease or neurological or psychiatric disorder that could influence quality of life measurement; inability to perform neuropsycological tests.

Ages: 33 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
work stress | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania, Catania, Italy